CLINICAL TRIAL: NCT04932070
Title: Berberine is an Effective Insulin Sensitizer and Improves Homeostasis of Metabolic and Hormonal Disorders in Women With Polycystic Ovary Syndrome: a Novel Treatment Strategy for PCOS
Brief Title: Berberine and Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1206/14122018
Record Dates: First submitted 2021-06-14; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Polycystic Ovary Syndrome; Berberine
Keywords: berberine; Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Berberine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Berberine (Experimental): 2 daily oral doses (one before lunch and one dinner) of 550 mg of berberine tablets
  Interventions: Dietary Supplement: Berberine

INTERVENTIONS:
Dietary Supplement: Berberine — 2 daily oral doses (one before lunch and one dinner) of 550 mg of berberine tablets

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is the most frequent endocrine disease in female reproductive-age. Recently, increasing evidence has shown that natural plant-based products may play a role in PCOS management. Previous study in PCOS preclinical model and in humans demonstrated that berberine is an effective insulin sensitizer and improves homeostasis of metabolic, inflammatory and hormonal disorders. However, to date there is no clinical study that considers globally all the activities carried out by berberine in PCOS clinical features. Given this background, aim of this study was to evaluate in normal-overweight PCOS women with normal menses the berberine effectiveness on: insulin resistance by Homeostasis Model Assessment (HOMA); inflammation by C-Reactive Protein (CRP), TNF-alpha; lipid metabolism; sex hormone profile and symptoms correlated to hyperandrogenism, such as acne, by Global Acne Grading System (GAGS) and Cardiff Acne Disability Index (CADI); body composition by dual-energy X-ray absorptiometry. All these parameters were collected at baseline and 60 days after supplementation with a new bioavailable and safe berberine formulation. Finally, adverse effects were assessed by liver and kidney functions. To evaluate statistically significant pre- post-supplementation changes, fitted a linear mixed model for each investigated endpoint was performed.

ELIGIBILITY:
Inclusion Criteria:

* normal and overweight women (Body Mass Index (BMI) 25-30 kg/m2)
* newly detected Polycystic Ovary Syndrome

Exclusion Criteria:

* any concomitant medication
* presence of liver, renal and thyroid disease
* smoking
* drinking more than two standard alcoholic beverages/day (20 g of alcohol/day)

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-05 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2021-01-26 (Actual)

PRIMARY OUTCOMES:
Changes on insulin resistance | Changes from baseline insulin resistance at 8 weeks
  Homeostasis Model Assessment (pt), for evaluate insulin resistance if > 2.4

SECONDARY OUTCOMES:
Changes on inflammation | Changes from baseline inflammation at 8 weeks
  C-Reactive Protein (mg/dl)
Changes on inflammation | Changes from baseline inflammation at 8 weeks
  Tumor Necrosis Factor alpha (pg/ml)
Changes on lipid profile | Changes from baseline lipid profile at 8 weeks
  Total Cholesterol (mg/dl), High Density Lipoprotein Cholesterol (mg/dl), Low Density Lipoprotein Cholesterol (mg/dl), Very Low Density Lipoprotein (mg/dl),Triglycerides (mg/dl)
Changes on Carbohydrate profile | Changes from baseline Carbohydrate profile at 8 weeks
  Glycemia (mg/dl)
Changes on Carbohydrate profile | Changes from baseline Carbohydrate profile at 8 weeks
  Insulin (mcU/ml)
Changes on Hormonal profile | Changes from baseline Hormonal profile at 8 weeks
  Sex Hormone Binding Globulin (nmol/l)
Changes on Hormonal profile | Changes from baseline Hormonal profile at 8 weeks
  Testosterone (ng/ml)
Changes on Hormonal profile | Changes from baseline Hormonal profile at 8 weeks
  Free Androgen Index (ratio)
Changes on safety | Changes from baseline safety at 8 weeks
  Aspartate aminotransferase (IU/l), alanine aminotransferase (IU/l)
Changes on safety | Changes from baseline safety at 8 weeks
  Total bilirubin (mg/dl)
Changes on safety | Changes from baseline safety at 8 weeks
  Gamma Glutamyl Transferase (U/I), Creatine Phosphokinase (U/I)
Changes on anthropometry | Changes from baseline anthropometry at 8 weeks
  waist circumference (cm), hip circumference (cm)
Changes on anthropometry | Changes from baseline anthropometry at 8 weeks
  Weight (kg)
Changes on anthropometry | Changes from baseline anthropometry at 8 weeks
  Body Mass Index (Kg/m2)
Changes on body composition | Changes from baseline body composition at 8 weeks
  Fat mass (g), lean mass (g), visceral adipose tissue (g)
Changes on acne assessment | Changes from baseline acne assessment at 8 weeks
  Global Acne Grading System (scale): each type of acne lesion is given a value depending on severity: no lesions = 0, comedones = 1, papules = 2, pustules = 3, and nodules = 4. Each of the location was graded separately on 0-4 scale, with the most severe lesion within that location determining the local score. The severity was then graded according to the global score which is the summation of all local scores. A score of 1-6 was considered mild; 7-18, moderate; 19- 26, severe; and 27-32, very severe. The maximum score was 32
Changes on acne assessment | Changes from baseline acne assessment at 8 weeks
  Cardiff Acne Disability Index (scale): the Cardiff Acne Disability Index consists of five questions with a Likert scale, four response categories (0-3). The five questions relate to feeling of aggression, frustration, interference with social life, avoidance of public changing facilities and appearance of the skin-all over the last month-and an indication of how bad the acne was now. The CADI score was calculated by summing the score of each question resulting in a possible maximum of 15 and minimum of 0. CADI scores were graded as low (0-4), medium (5-9), and high (10-15)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda di Servizi alla Persona, Pavia, Italy